CLINICAL TRIAL: NCT01251913
Title: A Pilot Study of Inpatient Hospice With Procurement of Brain Tumor Tissue on Expiration for Research Purposes
Status: Terminated | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110036; 11-C-0036
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2015-04-29

CONDITIONS: Ependymomas; Gliomas; PNET; Pineal Tumors; PCNSL (Primary CNS Lymphoma)
Keywords: Tissue Harvest; Hospice; Autopsy; Crainiotomy; Brain Tumor; Glioma; Astrocytoma
MeSH Terms: conditions — Ependymoma; Glioma; Neuroectodermal Tumors, Primitive; Pinealoma; Brain Neoplasms; Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- An important new area of brain tumor research is the development of tumor and brain stem cell lines. Successful growth of these cell lines requires obtaining large volumes of fresh tumor and brain tissue, which is best accomplished by harvesting whole brains from recently deceased patients. These cell lines will help researchers understand how these tumors develop and will also help identify new targets for treatment. Researchers are interested in conducting a pilot study of planned inpatient hospice care with timely brain tumor tissue harvest at the time of death.

Objectives:

* To provide high-quality end of life inpatient hospice care for patients with untreatable brain tumors.
* To procure brain and tumor tissue shortly after time of death in order to derive viable tumor and neural stem cell lines for research purposes.

Eligibility:

* Individuals at least 18 years of age who have an untreatable primary brain or central nervous system tumor, are able to give informed consent (either their own or through a designated power of attorney), and have agreed to a Do Not Resuscitate order and Consent for Autopsy as part of the end-of-life care plan.
* HIV-positive individuals or those suspected of having infectious cerebritis are not eligible because of the potential for contamination of brain tissue.

Design:

* Participants will be enrolled in inpatient hospice admission to the National Institutes of Health Clinical Center either from home or from an outside hospital once a study investigator estimates an expected survival of less than 2 weeks.
* Participants will receive palliative care at the Clinical Center. Care will be tailored to each participant depending on the information provided in the individual's end-of-life care plan.
* Supportive medications such as antiseizure medications and pain relievers will be administered as appropriate.
* At the time of death, researchers will follow standard procedures for notifying next of kin and will collect brain tissue and tumor samples from the deceased.
* Following tissue collection, the deceased will be released for autopsy and funeral procedures.

DETAILED DESCRIPTION:
BACKGROUND:

- Patients treated by the Neuro-Oncology Branch (NOB) for their brain tumors unfortunately and commonly succumb to their disease. They and their loved ones often seek a way of adding meaning and utility to their death by agreeing to donate brain tumor tissue for laboratory research that may serve the medical community, and ultimately other patients, through better understanding of these rare diseases. Important new avenues of brain tumor research includes the molecular characterization of tumor tissue, and the development of tumor and neural stem cell lines. Successful growth of these cell lines requires acquisition of large volumes of fresh tumor and brain tissue that can best be accomplished by harvesting whole brains from recently deceased patients. In an effort to provide high quality end of life care, with the additional intent of facilitating efficient donation of brain tumor tissue at the time of death, we are conducting a pilot study of planned inpatient hospice care incorporating timely brain tumor tissue procurement at the time of expiration.

OBJECTIVES:

* Provide high quality end of life inpatient hospice care for patients dying with untreatable brain tumors.
* Procure brain and tumor tissue shortly after time of death in order to derive viable tumor and neural stem cell lines for research purposes.

ELIGIBILITY:

- Adult patients with primary brain tumors.

DESIGN:

- This is a pilot study to assess feasibility of procuring viable brain and tumor tissue proximal to the time of death. Target accrual is 10 patients for brain harvest.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients with primary brain tumors including glioblastoma multiforme (GBM), gliosarcoma (GS), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), low grade astrocytoma, low grade oligoastrocytoma, low grade oligodendroglioma, astrocytoma NOS (not otherwise specified), radiographically diagnosed brain stem gliomas, primitive neuroectodermal tumors (PNETs, including medulloblastomas, supratentorial PNET), pineal tumors, glioneuronal tumors, ependymomas and primary central nervous system lymphomas.
  2. All patients or their LAR (Legally Authorized Individual) (if the patient is deemed by the treating physician to be impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study.
  3. Patients or their LAR and their legal next of kin must agree to a Do Not Resuscitate order and Consent for Autopsy as part of the end-of-life care plan.
  4. Patients must be greater than or equal to 18 years old, and with a life expectancy < two weeks.
  5. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.

EXCLUSION CRITERIA:

1. Known to be pregnant (known positive pregnancy test although such testing is not a requirement for enrollment).
2. HIV-positive patients or those suspected of infectious cerebritis/abscess are ineligible because of the potential for contamination of brain tissue.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-11-12; Study Completion 2015-04-29

PRIMARY OUTCOMES:
Provide high quality end of life inpatient hospice care for patients dying with untreatable brain tumors.

SECONDARY OUTCOMES:
Procure brain and tumor tissue shortly after time of death in order to derive viable tumor and neural stem cell lines for research purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Warren, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Deschavanne PJ, Fertil B. A review of human cell radiosensitivity in vitro. Int J Radiat Oncol Biol Phys. 1996 Jan 1;34(1):251-66. doi: 10.1016/0360-3016(95)02029-2. PMID 12118559
- [Background] Hecht BK, Turc-Carel C, Chatel M, Grellier P, Gioanni J, Attias R, Gaudray P, Hecht F. Cytogenetics of malignant gliomas: I. The autosomes with reference to rearrangements. Cancer Genet Cytogenet. 1995 Oct 1;84(1):1-8. doi: 10.1016/0165-4608(95)00091-7. PMID 7497435
- [Background] Pardal R, Clarke MF, Morrison SJ. Applying the principles of stem-cell biology to cancer. Nat Rev Cancer. 2003 Dec;3(12):895-902. doi: 10.1038/nrc1232. No abstract available. PMID 14737120